CLINICAL TRIAL: NCT04742764
Title: Dosing of Extracorporeal Cytokine Removal In Septic Shock (DECRISS): a Prospective, Randomized, Multicenter Clinical Trial
Brief Title: Extracorporal Cytokin Removal in Septic Shock: a Prospective, Randomized, Multicenter Clinical Trial
Acronym: DECRISS
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The human resources required to start enrollment were not available anymore.
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OGYÉI/65049/2020
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Septic Shock
Keywords: sepsis, septic shock, cytosorb, cytokine removal
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, three-arm, open-label, international, multi-centre, phase III study
Who Masked: Outcomes Assessor
Masking Description: No masking is applied in this study, as it is impossible to blind the medical personnel and participants. Statisticians will be blinded to allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Patients randomized to standard medical therapy.
  Interventions: Combination Product: Standard medical therapy
- Group B (Active Comparator): Patients randomized to cytokine removal therapy with Cytosorb, with the adsorber device changed in every 12 hours.
  Interventions: Device: Standard medical therapy plus cytokine removal treatment using Cytosorb, with the adsorber changed in every 12 hours
- Group C (Active Comparator): Patients randomized to cytokine removal therapy with Cytosorb, with the adsorber device changed in every 24 hours.
  Interventions: Device: Standard medical therapy plus cytokine removal treatment using Cytosorb, with the adsorber changed in every 24 hours

INTERVENTIONS:
Combination Product: Standard medical therapy — Standard medical therapy (according to the Surviving Sepsis Campaign) will include standard monitoring (pulseoximetry, 5-lead ECG, continuous invasive blood pressure monitoring, central venous cannulation and 24 with PiCCO-technology. Norepinephrine as a vasopressor and dobutamine - if needed - as an inotrope will be administered by the attending physician.
  Arms: Group A
Device: Standard medical therapy plus cytokine removal treatment using Cytosorb, with the adsorber changed in every 12 hours — Standard medical therapy, as discussed above will be applied. Furthermore, Cytosorb will be administered as soon as it is possible after randomization but not later than 2 hour (start of the treatment, T0). In a blood pump circuit in pre-haemofilter position, using a kidney replacement device of Fresenius Multifiltrate as a solo therapy or in combination with renal replacement therapy. It will be run in CVVHD, CVVHDF or CVVH mode with a 150 and 200 ml/min blood flow. Anticoagulation will be applied intravenously with heparin, low molecular weight heparin or citrate. The aim of the pump flow rate will be 100-400 mL/min, and the flow rate will be recorded. Possible shock reversal will be assessed by the physician attending. Adsorber cartridges will be changed in every 12 hours. End of the study period (Te): 12 hours after shock reversal, death of the patient, or maximum of five days, whichever happens first.
  Arms: Group B
Device: Standard medical therapy plus cytokine removal treatment using Cytosorb, with the adsorber changed in every 24 hours — The standard medical therapy and method of Cytosorb treatment as detailed above will be applied. Adsorber cartridges will be changed in every 24 hours.
  Arms: Group C

SUMMARY:
Sepsis and septic shock have mortality rates between 20-50%. When standard therapeutic measures fail to improve patients' condition, additional therapeutic alternatives are applied to reduce morbidity and mortality. One of the most recent alternatives is extracorporeal cytokine hemoadsorption. One of the most tested devices is CytoSorb, however, there are a lot of open questions, such timing, dosing and of course its overall efficacy. This study aims to compare the efficacy of standard medical therapy (Group A, SMT) and continuous extracorporeal cytokine removal with CytoSorb therapy in patients with early refractory septic shock. Furthermore, we compare the dosing of CytoSorb adsorber device - as the cartridge will be changed in every (12 Group B) or 24 hours (Group C).

ELIGIBILITY:
Inclusion Criteria:

* Septic shock as defined by the Sepsis-3 criteria
* Septic shock both medical or surgical ethiology (except for re-operation)
* APACHE > 25
* Mechanical ventilation
* Norepinephrine requirement ≥0.4 µg/kg/min for at least 30 minutes, when hypovolemia is highly unlikely as indicated by invasive hemodynamic measurements assessed by the attending physician
* Invasive hemodynamic monitoring to determine cardiac output and derived variables
* Procalcitonin level ≥ 10 ng/ml
* Inclusion within 6 - 24 hours after the onset of vasopressor need and after all standard therapeutic measures have been implemented without clinical improvement (i.e.: the shock is considered refractory)

Exclusion Criteria:

* Patients under 18 years and over 80
* Lack of health insurance
* Pregnancy
* Standard guideline-based medical treatment not exhausted (detailed below at 3.6) standard medical therapy)
* End stage organ failure
* New York Heart Association Class IV.
* Chronic renal failure with eGFR < 15 ml/min/1,73 m2
* End-stage liver disease (MELD score >30, Child-Pugh score Class C
* Unlikely survival for 24 hours according to the attending physician
* Acute onset of hemato-oncological illness
* Post cardiopulmonary resuscitation care
* Re-operation in context with the septic insult
* Immunosuppression
* systemic steroid therapy (>10 mg prednisolon/day)
* immunosuppressive agents (i.e.: methotrexate, azathioprine, cyclosporin, tacrolimus, cyclophosphamide)
* Human immunodeficiency virus infection (active AIDS): HIV-VL > 50 copies/mL
* Patients with transplanted vital organs
* Thrombocytopenia (<20.000/ml)
* More than 10%-of body surface area with a third-degree burn
* Acute coronary syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Shock reversal | At the time of shock reversal assessed up to 5 days
  Proportion of patients achieving shock reversal, defined as follows:
  no need (or minimal need, meaning max. the 10% of the maximum dose) of vasopressore for 3 hours, with haemodynamic measurements, and arterial, central venous blood gas analysis, arterial lactate level measurement, venous and arterial pCO2-gap and O2 saturation measurements to confirm cardiorespiratory stability
Time to shock reversal | From the start of the treatment until shock reversal assessed up to 5 days
  The time from the start of the treatment (T0) until shock reversal

SECONDARY OUTCOMES:
Procalcitonine level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of procalcitonine
Change in procalcitonine level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in procalcitonine level from the start of the treatment until the end of the study period
Interleukin-6 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of interleukin-6
Change in interleukin-6 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in interleukin-6 level from the start of the treatment until the end of the study period
C-reactive protein level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of C-reactive protein
Change in C-reactive protein level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in C-reactive protein level from the start of the treatment until the end of the study period
Interleukin-1 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of interleukin-1
Change in interleukin-1 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in interleukin-1 level from the start of the treatment until the end of the study period
Interleukin-1ra level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of interleukin-1ra
Change in interleukin-1ra level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in interleukin-1ra level from the start of the treatment until the end of the study period
Interleukin-8 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of interleukin-8
Change in interleukin-8 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in interleukin-8 level from the start of the treatment until the end of the study period
Interleukin-10 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of interleukin-10
Change in interleukin-10 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in interleukin-10 level from the start of the treatment until the end of the study period
Tumor necrosis factor alpha level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of tumor necrosis factor alpha
Change in tumor necrosis factor alpha level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in tumor necrosis factor alpha level from the start of the treatment until the end of the study period
Syndecan-1 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of syndecan-1
Change in syndecan-1 level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in syndecan-1 level from the start of the treatment until the end of the study period
Heparan sulphate level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of heparan sulphate
Change in heparan sulphate level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in heparan sulphate level from the start of the treatment until the end of the study period
Arterial lactate levels | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Absolute level of arterial lactate levels
Change in arterial lactate levels level | 0, 6, 12,24 hours after the start of the treatment, then daily until the end of study period assessed up to 90 +/- 7 days at second follow-up visit
  Change in arterial lactate level from the start of the treatment until the end of the study period
Change in SOFA score | From the start of the treatment until the end of the treatment assessed up to 5 days
  Change in SOFA score from the start of the treatment until the end of the study period
Change in extravascular lung water (EVLW) | From the start of the treatment until the end of the treatment assessed up to 5 days
  Change in extravascular lung water (EVLW) from the start of the treatment until the end of the study period
Duration of mechanical ventilation | From the start of the treatment until the end of the treatment assessed up to 5 days
  Duration of mechanical ventilation given in days
Duration of catecholamine requirement | From the start of the catecholamine requirement until the end of the catecholamine requirement assessed up to 5 days
  Duration of catecholamine requirement given in days
Duration of renal replacement therapy | From the start of the renal replacement therapy requirement until the end of the renal replacement therapy requirement assessed up to 90+/-7 days at the second follow-up visit
  Duration of renal replacement therapy given in days
Need for dialysis | day 28±7, day 90±7
  Rate of patients, who require dialysis
Length of internsive care unit stay | From admission to intensive care unit until the end of intensive care unit assessed at study completion an avarage of 90 days
  Length of intensive care unit stay given in days
Length of hospital stay | From admission to the hospital until the end of hospital stay assessed at study completion an avarage of 90 days
  Length of hospital stay given in days
Survival | Rate if surviving patients assessed at death, or study completion which ever happens first, up to 90 +/-7 days
  Rate of surviving patients
Adverse events | Recorded at the occurrance of adverse events, and study completion up to 90 +/- 7 days
  Rate of patients experiencing adverse events, or device deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: Péter Hegyi, MD, PhD, DSc, Principal Investigator — Insitute for Translational Medicine, University of Pécs, Medical School, Pécs, Hungary
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sogayar AM, Machado FR, Rea-Neto A, Dornas A, Grion CM, Lobo SM, Tura BR, Silva CL, Cal RG, Beer I, Michels V, Safi J, Kayath M, Silva E; Costs Study Group - Latin American Sepsis Institute. A multicentre, prospective study to evaluate costs of septic patients in Brazilian intensive care units. Pharmacoeconomics. 2008;26(5):425-34. doi: 10.2165/00019053-200826050-00006. PMID 18429658
- [Background] Adrie C, Alberti C, Chaix-Couturier C, Azoulay E, De Lassence A, Cohen Y, Meshaka P, Cheval C, Thuong M, Troche G, Garrouste-Orgeas M, Timsit JF. Epidemiology and economic evaluation of severe sepsis in France: age, severity, infection site, and place of acquisition (community, hospital, or intensive care unit) as determinants of workload and cost. J Crit Care. 2005 Mar;20(1):46-58. doi: 10.1016/j.jcrc.2004.10.005. PMID 16015516
- [Background] Khwannimit B, Bhurayanontachai R. The direct costs of intensive care management and risk factors for financial burden of patients with severe sepsis and septic shock. J Crit Care. 2015 Oct;30(5):929-34. doi: 10.1016/j.jcrc.2015.05.011. Epub 2015 May 20. PMID 26051981
- [Background] Iskander KN, Osuchowski MF, Stearns-Kurosawa DJ, Kurosawa S, Stepien D, Valentine C, Remick DG. Sepsis: multiple abnormalities, heterogeneous responses, and evolving understanding. Physiol Rev. 2013 Jul;93(3):1247-88. doi: 10.1152/physrev.00037.2012. PMID 23899564
- [Background] Kwan A, Hubank M, Rashid A, Klein N, Peters MJ. Transcriptional instability during evolving sepsis may limit biomarker based risk stratification. PLoS One. 2013;8(3):e60501. doi: 10.1371/journal.pone.0060501. Epub 2013 Mar 27. PMID 23544148
- [Background] Akira S, Uematsu S, Takeuchi O. Pathogen recognition and innate immunity. Cell. 2006 Feb 24;124(4):783-801. doi: 10.1016/j.cell.2006.02.015. PMID 16497588
- [Background] Hotchkiss RS, Monneret G, Payen D. Sepsis-induced immunosuppression: from cellular dysfunctions to immunotherapy. Nat Rev Immunol. 2013 Dec;13(12):862-74. doi: 10.1038/nri3552. Epub 2013 Nov 15. PMID 24232462
- [Background] Schulte W, Bernhagen J, Bucala R. Cytokines in sepsis: potent immunoregulators and potential therapeutic targets--an updated view. Mediators Inflamm. 2013;2013:165974. doi: 10.1155/2013/165974. Epub 2013 Jun 18. PMID 23853427
- [Background] Venet F, Lukaszewicz AC, Payen D, Hotchkiss R, Monneret G. Monitoring the immune response in sepsis: a rational approach to administration of immunoadjuvant therapies. Curr Opin Immunol. 2013 Aug;25(4):477-83. doi: 10.1016/j.coi.2013.05.006. Epub 2013 May 28. PMID 23725873
- [Background] Sharawy N. Vasoplegia in septic shock: do we really fight the right enemy? J Crit Care. 2014 Feb;29(1):83-7. doi: 10.1016/j.jcrc.2013.08.021. Epub 2013 Oct 4. PMID 24095623
- [Background] Laszlo I, Trasy D, Molnar Z, Fazakas J. Sepsis: From Pathophysiology to Individualized Patient Care. J Immunol Res. 2015;2015:510436. doi: 10.1155/2015/510436. Epub 2015 Jul 15. PMID 26258150
- [Background] Bellomo R, Baldwin I, Ronco C. Extracorporeal blood purification therapy for sepsis and systemic inflammation: its biological rationale. Contrib Nephrol. 2001;(132):367-74. doi: 10.1159/000060105. PMID 11395904
- [Background] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Background] Kreymann KG, de Heer G, Nierhaus A, Kluge S. Use of polyclonal immunoglobulins as adjunctive therapy for sepsis or septic shock. Crit Care Med. 2007 Dec;35(12):2677-85. PMID 18074464
- [Background] Basu R, Pathak S, Goyal J, Chaudhry R, Goel RB, Barwal A. Use of a novel hemoadsorption device for cytokine removal as adjuvant therapy in a patient with septic shock with multi-organ dysfunction: A case study. Indian J Crit Care Med. 2014 Dec;18(12):822-4. doi: 10.4103/0972-5229.146321. PMID 25538418
- [Background] Bedina, E., et al., Hemoadsorption by cytosorb® in septic shock with acute kidney injury: A case series. Blood Purification, 2018. 46(3): p. 183-184.
- [Background] Bracht, H., et al., Pattern of cytokine removal using an adsorption column CytoSorb® during severe Candia albicans induced septic shock. Infection, Supplement, 2013. 41(1): p. S64-S65.
- [Background] Kellum JA, Venkataraman R, Powner D, Elder M, Hergenroeder G, Carter M. Feasibility study of cytokine removal by hemoadsorption in brain-dead humans. Crit Care Med. 2008 Jan;36(1):268-72. doi: 10.1097/01.CCM.0000291646.34815.BB. PMID 18090355
- [Background] Namas RA, Namas R, Lagoa C, Barclay D, Mi Q, Zamora R, Peng Z, Wen X, Fedorchak MV, Valenti IE, Federspiel WJ, Kellum JA, Vodovotz Y. Hemoadsorption reprograms inflammation in experimental gram-negative septic peritonitis: insights from in vivo and in silico studies. Mol Med. 2012 Dec 20;18(1):1366-74. doi: 10.2119/molmed.2012.00106. PMID 22751621
- [Background] Peng ZY, Carter MJ, Kellum JA. Effects of hemoadsorption on cytokine removal and short-term survival in septic rats. Crit Care Med. 2008 May;36(5):1573-7. doi: 10.1097/CCM.0b013e318170b9a7. PMID 18434884
- [Background] Peng ZY, Wang HZ, Carter MJ, Dileo MV, Bishop JV, Zhou FH, Wen XY, Rimmele T, Singbartl K, Federspiel WJ, Clermont G, Kellum JA. Acute removal of common sepsis mediators does not explain the effects of extracorporeal blood purification in experimental sepsis. Kidney Int. 2012 Feb;81(4):363-9. doi: 10.1038/ki.2011.320. Epub 2011 Sep 14. PMID 21918497
- [Background] Friesecke S, Trager K, Schittek GA, Molnar Z, Bach F, Kogelmann K, Bogdanski R, Weyland A, Nierhaus A, Nestler F, Olboeter D, Tomescu D, Jacob D, Haake H, Grigoryev E, Nitsch M, Baumann A, Quintel M, Schott M, Kielstein JT, Meier-Hellmann A, Born F, Schumacher U, Singer M, Kellum J, Brunkhorst FM. International registry on the use of the CytoSorb(R) adsorber in ICU patients : Study protocol and preliminary results. Med Klin Intensivmed Notfmed. 2019 Nov;114(8):699-707. doi: 10.1007/s00063-017-0342-5. Epub 2017 Sep 4. PMID 28871441
- [Background] Friesecke S, Stecher SS, Gross S, Felix SB, Nierhaus A. Extracorporeal cytokine elimination as rescue therapy in refractory septic shock: a prospective single-center study. J Artif Organs. 2017 Sep;20(3):252-259. doi: 10.1007/s10047-017-0967-4. Epub 2017 Jun 6. PMID 28589286
- [Background] Kogelmann K, Jarczak D, Scheller M, Druner M. Hemoadsorption by CytoSorb in septic patients: a case series. Crit Care. 2017 Mar 27;21(1):74. doi: 10.1186/s13054-017-1662-9. PMID 28343448
- [Background] Hawchar F, Laszlo I, Oveges N, Trasy D, Ondrik Z, Molnar Z. Extracorporeal cytokine adsorption in septic shock: A proof of concept randomized, controlled pilot study. J Crit Care. 2019 Feb;49:172-178. doi: 10.1016/j.jcrc.2018.11.003. Epub 2018 Nov 10. PMID 30448517
- [Background] Brouwer WP, Duran S, Kuijper M, Ince C. Hemoadsorption with CytoSorb shows a decreased observed versus expected 28-day all-cause mortality in ICU patients with septic shock: a propensity-score-weighted retrospective study. Crit Care. 2019 Sep 18;23(1):317. doi: 10.1186/s13054-019-2588-1. PMID 31533846
- [Background] Öveges N, L.s.I., Forgács M, et al, Procalcitonin elimination during cytokine adsorption therapy in septic shock: a spin-off study of the ACESS trial. Crit Care, 2017. 21:383.
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Amendola A, Sberna G, Forbici F, Abbate I, Lorenzini P, Pinnetti C, Antinori A, Capobianchi MR. The dual-target approach in viral HIV-1 viremia testing: An added value to virological monitoring? PLoS One. 2020 Feb 5;15(2):e0228192. doi: 10.1371/journal.pone.0228192. eCollection 2020. PMID 32023284
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Kogelmann K, Scheller M, Druner M, Jarczak D. Use of hemoadsorption in sepsis-associated ECMO-dependent severe ARDS: A case series. J Intensive Care Soc. 2020 May;21(2):183-190. doi: 10.1177/1751143718818992. Epub 2019 Jan 8. PMID 32489416
- [Background] Wani SJ, Mufti SA, Jan RA, Shah SU, Qadri SM, Khan UH, Bagdadi F, Mehfooz N, Koul PA. Combination of vitamin C, thiamine and hydrocortisone added to standard treatment in the management of sepsis: results from an open label randomised controlled clinical trial and a review of the literature. Infect Dis (Lond). 2020 Apr;52(4):271-278. doi: 10.1080/23744235.2020.1718200. Epub 2020 Jan 28. PMID 31990246
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Peake SL, Bailey M, Bellomo R, Cameron PA, Cross A, Delaney A, Finfer S, Higgins A, Jones DA, Myburgh JA, Syres GA, Webb SA, Williams P; ARISE Investigators, for the Australian and New Zealand Intensive Care Society Clinical Trials Group. Australasian resuscitation of sepsis evaluation (ARISE): A multi-centre, prospective, inception cohort study. Resuscitation. 2009 Jul;80(7):811-8. doi: 10.1016/j.resuscitation.2009.03.008. Epub 2009 May 20. PMID 19467755
- [Background] Girbes ARJ, de Grooth HJ. Time to stop randomized and large pragmatic trials for intensive care medicine syndromes: the case of sepsis and acute respiratory distress syndrome. J Thorac Dis. 2020 Feb;12(Suppl 1):S101-S109. doi: 10.21037/jtd.2019.10.36. PMID 32148932
- [Background] Vincent JL. We should abandon randomized controlled trials in the intensive care unit. Crit Care Med. 2010 Oct;38(10 Suppl):S534-8. doi: 10.1097/CCM.0b013e3181f208ac. PMID 21164394
- [Background] Jozwiak M, Teboul JL, Monnet X. Extravascular lung water in critical care: recent advances and clinical applications. Ann Intensive Care. 2015 Dec;5(1):38. doi: 10.1186/s13613-015-0081-9. Epub 2015 Nov 6. PMID 26546321
- [Background] David S, Thamm K, Schmidt BMW, Falk CS, Kielstein JT. Effect of extracorporeal cytokine removal on vascular barrier function in a septic shock patient. J Intensive Care. 2017 Jan 21;5:12. doi: 10.1186/s40560-017-0208-1. eCollection 2017. PMID 28127437
- [Background] Riedel S. Procalcitonin and the role of biomarkers in the diagnosis and management of sepsis. Diagn Microbiol Infect Dis. 2012 Jul;73(3):221-7. doi: 10.1016/j.diagmicrobio.2012.05.002. PMID 22704255
- [Background] Nylen ES, Whang KT, Snider RH Jr, Steinwald PM, White JC, Becker KL. Mortality is increased by procalcitonin and decreased by an antiserum reactive to procalcitonin in experimental sepsis. Crit Care Med. 1998 Jun;26(6):1001-6. doi: 10.1097/00003246-199806000-00015. PMID 9635646
- [Background] Schadler D, Pausch C, Heise D, Meier-Hellmann A, Brederlau J, Weiler N, Marx G, Putensen C, Spies C, Jorres A, Quintel M, Engel C, Kellum JA, Kuhlmann MK. The effect of a novel extracorporeal cytokine hemoadsorption device on IL-6 elimination in septic patients: A randomized controlled trial. PLoS One. 2017 Oct 30;12(10):e0187015. doi: 10.1371/journal.pone.0187015. eCollection 2017. PMID 29084247
- [Background] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Laszlo I, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z; EProK study group. Early procalcitonin kinetics and appropriateness of empirical antimicrobial therapy in critically ill patients: A prospective observational study. J Crit Care. 2016 Aug;34:50-5. doi: 10.1016/j.jcrc.2016.04.007. Epub 2016 Apr 13. PMID 27288610
- [Derived] Kanjo A, Molnar Z, Zadori N, Gede N, Eross B, Szako L, Kiss T, Marton Z, Malbrain MLNG, Szuldrzynski K, Szrama J, Kusza K, Kogelmann K, Hegyi P. Dosing of Extracorporeal Cytokine Removal In Septic Shock (DECRISS): protocol of a prospective, randomised, adaptive, multicentre clinical trial. BMJ Open. 2021 Aug 26;11(8):e050464. doi: 10.1136/bmjopen-2021-050464. PMID 34446497